CLINICAL TRIAL: NCT05138978
Title: Metagenomic and Metatranscriptomic Analysis of Clinical Plaque Samples
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: ERO-2015-PLA-07-RPS
Record Dates: First submitted 2021-11-16; First posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Plaque
MeSH Terms: conditions — Plaque, Amyloid

STUDY DESIGN:
Intervention Model Description: Each subject will be randomized.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colgate Maximum Cavity Protection plus Sugar Acid Neutralizer (Experimental): Toothpaste
  Interventions: Drug: Colgate Maximum Cavity Protection plus Sugar Acid Neutralizer
- Colgate Cavity Protection (Other): Toothpaste
  Interventions: Drug: Colgate Cavity Protection

INTERVENTIONS:
Drug: Colgate Maximum Cavity Protection plus Sugar Acid Neutralizer — Toothpaste
  Arms: Colgate Maximum Cavity Protection plus Sugar Acid Neutralizer
Drug: Colgate Cavity Protection — Toothpaste
  Arms: Colgate Cavity Protection

SUMMARY:
The objective of this study is to determine the metagenomic and metatranscriptomic analysis of clinical samples.

DETAILED DESCRIPTION:
This study is a blinded, non-randomized, crossover design. Subjects who meet the inclusion/exclusion criteria will be enrolled in the study. Following enrollment, subjects will be asked to use a washout dentifrice (#200000035883/001/000) for a minimum of 1 week. Fasting plaque will be collected at Baseline and then again at a duplicate baseline collection up to 1 week after the baseline collection. Subjects will be assigned a new dentifrice (#200000035883/001/000) to use for 12 weeks. After 12 weeks' use, fasting plaque will be collected. There will be a duplicate plaque collection up to 1 week after 12 week collection. Subjects will be given a new dentifrice (#200000040228/001/000) to use for the next 24 weeks. After 24 weeks' use, fasting plaque will be collected, and there will be a duplicate plaque collection up to 1 week after this collection.

ELIGIBILITY:
Inclusion Criteria

* Male and/or female subjects 16 years and above
* Minimum of 20 natural uncrowned teeth (excluding third molars) must be present
* Caries active subjects will have at least 3 active caries lesions (ICDAS score 1 - 3). Caries free control subjects will either have ICDAS score 0 or ICDAS score of 1 - 3 where the lesion is inactive.
* Available throughout entire study
* Willing to use only assigned products for oral hygiene throughout the duration of the study
* Must give written informed consent
* Must be in good general health

Exclusion Criteria

* Unwilling or unable to sign an Informed Consent Form
* Advanced periodontal disease
* Medical condition which requires premedication prior to dental visits/procedures
* Diseases of the soft or hard oral tissues
* Orthodontic appliances that interfere with clinical assessments
* Impaired salivary function
* Current use of drugs that can affect salivary flow
* Use antibiotics 3 months prior to or during this study
* Use of any arginine containing oral care products such as Colgate Sensitive Pro-Relief and Colgate Maximum Cavity Protection plus Sugar Acid Neutralizer dentifrices 3 months prior to or during this study
* Pregnant or breastfeeding
* Participate in another clinical study 1 week prior to the start of the washout period or during the study period
* Use of tobacco products
* Allergic to common dentifrice ingredients
* Allergic to amino acids
* Immune compromised individuals (HIV, AIDS, immuno-suppressive drug therapy)

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-10-06 (Actual); Primary Completion 2018-10-17 (Actual); Study Completion 2018-10-17 (Actual)

PRIMARY OUTCOMES:
DNA (metagenomic) sequences | 38 weeks
  The primary outcome is to collect plaque following each treatment and to assess DNA
RNA (metatranscriptomic) sequences | 38 weeks
  The primary outcome is to collect plaque following each treatment and to assess RNA

CONTACTS AND LOCATIONS:
Overall Officials: Luciana Rinaudi-Marron, DR, Study Director — Colgate Palmolive
Locations (1):
- King's College London Dental Institute, UK, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided